CLINICAL TRIAL: NCT01678781
Title: Open International Study on Quality of Life in IBS Patients Before and After 8 Weeks Treatment With Mebeverine/Pinaverium Bromide
Brief Title: Open International Study on Quality of Life in Irritable Bowel Syndrome (IBS) Patients Before and After 8 Weeks Treatment With Mebeverine/Pinaverium Bromide
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: CHILTERN International GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: P13-678
Record Dates: First submitted 2012-07-13; First posted 2012-09-05 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Abdominal pain; Diarrhea; Mebeverine hydrochloride; Constipation; Pinaverium bromide; Irritable bowel syndrome; Bloating; Quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Diarrhea; Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One patient group: Patients suffering from irritable bowel syndrome

SUMMARY:
A study to evaluate, by country and overall, the changes from baseline of the irritable bowel syndrome quality of life (IBS QoL) total score after 4 and 8 weeks of treatment with Duspatalin® or Dicetel® in IBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome patients diagnosed by Rome III criteria (18 years or older)

Exclusion Criteria:

* Pregnancy and lactation
* Specific contraindications to mebeverine hydrochloride or pinaverium bromide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 607 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Irritable Bowel syndrome (IBS) quality of life (QoL) measure (IBS-QoL) to assess the impairment of QoL in IBS patients | From baseline up to the week 8 visit

SECONDARY OUTCOMES:
Change in abdominal pain | From baseline up to the week 8 visit
Change in bloating | From baseline up to the week 8 visit
Change in feeling of abdominal distension | From baseline up to the week 8 visit
Change in stool frequency | From baseline up to the week 8 visit
Change in stool form | From baseline up to the week 8 visit
Change in straining of evacuation | From baseline up to the week 8 visit
Change in urgency of evacuation | From baseline up to the week 8 visit
Change in feeling of incomplete evacuation | From baseline up to the week 8 visit

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Krause, Study Director — Abbott
Locations (24):
- China (7):
  - Site reference ID/Investigator# 94519, Beijing
  - Site reference ID/Investigator# 94521, Guangzhou
  - Site reference ID/Investigator# 95475, Guangzhou
  - Site reference ID/Investigator # 94518, Shanghai
  - Site reference ID/Investigator # 94517, Shanghai
  - Site reference ID/Investigator # 94516, Shanghai
  - Site reference ID/Investigator # 94515, Wuhan
- Egypt (6):
  - Site Reference ID/Investigator# 95908, Alexandria
  - Site reference ID/Investigator# 95900, Cairo
  - Site reference ID/Investigator# 95901, El Sharkya
  - Site reference ID/Investigator# 95902, Giza
  - Site reference ID/Investigator# 95903, Giza
  - Site Reference ID/Investigator# 95906, Port Said
- Mexico (3):
  - Site reference ID/Investigaot# 94525, Guadalajara
  - Site refernce ID/Investigator# 94527, Mexico City
  - Site reference ID/Investigator# 94523, Tampico
- Poland (8):
  - Site reference ID/Investigator# 85314, Bialystok
  - Site Reference ID/Investigator# 85297, Bialystok
  - Site Reference ID/Investigator# 85298, Bydgoszcz
  - Site Reference ID/Investigator# 85293, Katowice
  - Site Reference ID/Investigator# 85296, Lodz
  - Site reference ID/Investigator# 85313, Olsztyn
  - Site Reference ID/Investigator# 85295, Poznan
  - Site Reference ID/Investigator# 85294, Poznan